CLINICAL TRIAL: NCT05755438
Title: A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream in Participants With Prurigo Nodularis
Brief Title: A Study to Evaluate the Safety and Efficacy of Ruxolitinib Cream in Participants With Prurigo Nodularis (PN)
Acronym: TRuE-PN1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB 18424-319; 2022-501621-20-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2023-01-25; First posted 2023-03-06 (Actual); Results first posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Prurigo
Keywords: Prurigo; Prurigo Nodularis; PN; Skin Diseases; Dermatitis; Eczematous; ruxolitinib; INCB 18424
MeSH Terms: conditions — Prurigo; Skin Diseases; Dermatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vehicle Cream BID (Placebo Comparator): Participants apply ruxolitinib matching vehicle cream topically to the affected areas as a thin film twice daily (BID) for 12 weeks during the DBVC period. Participants who have completed the treatment during DBVC period will apply ruxolitinib 1.5% cream topically during the open label extension (OLE) period for up to 40 weeks.
  Interventions: Drug: Vehicle Cream
- Ruxolitinib 1.5% Cream (Experimental): Participants apply ruxolitinib 1.5% cream topically to the affected areas as a thin film BID for 12 weeks during the DBVC period. Participants who have completed the treatment during DBVC period will apply ruxolitinib 1.5% cream the open label extension (OLE) period for up to 40 weeks.
  Interventions: Drug: Ruxolitinib Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream 1.5% twice daily (BID) during the vehicle controlled (DBVC)and open label treatment period (OLE).
  Other Names: INCB018424 phosphate cream
  Arms: Ruxolitinib 1.5% Cream
Drug: Vehicle Cream — Ruxolitinib matching vehicle cream 1.5% twice daily (BID) during the vehicle controlled period (DBVC).
  Arms: Vehicle Cream BID

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of Ruxolitinib cream in participants with Prurigo Nodularis (PN).

DETAILED DESCRIPTION:
The study comprises of a 12 week double-blind, vehicle-controlled (DBVC) treatment period, followed by a 40 week open label extension period, and 30 day safety follow-up period During the double blind period, all PN-affected areas identified at baseline will be treated, and during the open label period, only active PN-affected areas will be treated.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of PN ≥ 3 months before screening.
* ≥ 6 pruriginous lesions on ≥ 2 different body areas (such as right and left leg) at screening and baseline having a treatment area <20% BSA.
* IGA-CPG-S score of ≥ 2 at screening and baseline.
* Baseline PN-related WI-NRS score ≥ 7.
* Willingness to avoid pregnancy or fathering children.

Exclusion Criteria:

* Chronic pruritus due to a condition other than PN
* Total estimated BSA treatment area (excluding the scalp) > 20%.
* Neuropathic and psychogenic pruritus
* Active atopic dermatitis lesions within 3 months of screening and baseline.
* Uncontrolled thyroid function
* Concurrent skin or other serious or unstable medical conditions which may interfere with the evaluation of PN such as immunocompromised status, acute/chronic infections, active malignancy, history of TB, history of DVT/VTE, etc Protocol defined abnormal laboratory results.
* Use of any protocol-defined prohibited medication unless a washout is completed or use of medication known to cause itching.
* Psoralen and ultraviolet A or ultraviolet B therapy within 4 weeks before baseline or Ultraviolet light therapy or prolonged exposure to natural or artificial sources of ultraviolet radiation (within 2 weeks before baseline
* Pregnant or lactating, or considering pregnancy.
* History of alcoholism or drug addiction within 1 year
* Known allergy or reaction to any of the components of the study drug.
* Committed to a mental health institution by virtue of an order issued either by the judicial or the administrative authorities.
* Employees of the sponsor or investigator or otherwise dependents of them.
* The following participants are excluded in France:

  1. Vulnerable populations according to article L.1121-6 of the French Public Health Code.
  2. Adults under legal protection or who are unable to express their consent per article L.1121-8 of the French Public Health Code.
  3. Individuals not affiliated with the social security system.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-08-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haq Nawaz, md, Study Director — Incyte Corporation
Locations (71):
- United States (18):
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - Johnson Dermatology, Fort Smith, Arkansas
  - First Oc Dermatology, Fountain Valley, California
  - Dermatology Associates Pc, Rockville, Maryland
  - Clarkston Medical Group, Clarkston, Michigan
  - Revival Research Institute, Llc Troy, Troy, Michigan
  - Medisearch Clinical Trials, Saint Joseph, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - UC Health, Llc, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Central Sooner Research, Norman, Oklahoma
  - Dermatology Associates of Plymouth Meeting, Plymouth Meeting, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - International Clinical Research Tennessee Llc, Murfreesboro, Tennessee
  - North Texas Center For Clinical Research Ntccr, Frisco, Texas
  - Austin Institute For Clinical Research Aicr Pflugerville, Pflugerville, Texas
  - Center For Clinical Studies, Webster, Texas
  - Premier Clinical Research, Spokane, Washington
- Argentina (8):
  - Conexa Investigacion Clinica S.A., Buenos Aires
  - Cedic Centro de Investigaciones Clinicas, Ciudad Autonoma Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Psoriahue-Medicina Interdisciplinar, Ciudad Autonoma Buenos Aires
  - Centro de Investigaciones Medicas Mar Del Plata, Mar del Plata
  - Fundacion Scherbovsky, Mendoza
  - Instituto de Especialidades de La Salud Rosario, Rosario
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán
- Belgium (7):
  - Ulb Hospital Erasme, Brussels
  - Cliniques Universitaires Ucl Saint-Luc, Brussels
  - Az Sint-Lucas, Ghent
  - Universitair Ziekenhuis Gent, Ghent
  - Universitair Ziekenhuis (Uz) Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege - Sart Tilman, Liège
  - Chu Ucl Namur de Saint Elisabeth, Namur
- Canada (5):
  - Beacon Dermatology, Calgary, Alberta
  - Simcomed Health Ltd, Barrie, Ontario
  - Dermeffects, London, Ontario
  - Research Toronto, Toronto, Ontario
  - Centre de Recherche Saint-Louis, Québec, Quebec
- Chile (3):
  - Centro Medico Skinmed, Las Condes
  - Ciec - Centro Internacional de Estudios Cli-Nicos, Santiago
  - Clinical Research Chile Spa., Valdivia
- France (4):
  - Hospital Prive D'Antony, Antony
  - Hospital Morvan, Brest
  - Centre Hospitalier Universitaire de Nantes (Chu de Nantes) - Hotel-Dieu, Nantes
  - University Hospital of Saint Etienne, Saint-Etienne
- Germany (7):
  - University Medical Center Rwth Aachen, Aachen
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim
  - Universitaetsklinikum Carl Gustav Carus Tu Dresden, Dresden
  - Universitatsklinikum Schleswig Holstein, Kiel
  - Universitatsmedizin Der Johannes Gutenberg-Universitat Mainz Iii, Mainz
  - Universitats-Hautklink Tubingen, Tübingen
  - Hautarztpraxis Dr. Med. Matthias Hoffmann, Witten
- Italy (6):
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia (Presidio Spedali Civili), Brescia
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico San Marco, Catania
  - Asl 1 Avezzano L'Aquila Sulmona- Ospedale Regionale San Salvatore, Coppito
  - Azienda Ospedaliera Universitaria Policlinico 'Federico Ii', Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs, Roma
  - Ospedali Riuniti Di Ancona, Torrette
- Netherlands (2):
  - Amsterdam University Medical Centre, Amsterdam
  - Bravis Ziekenhuis, Bergen op Zoom
- Poland (6):
  - Pratia McM Krakow, Krakow
  - ETG LODZ, Lodz
  - Kliniczny Szpital Wojewodzki Nr 1, Rzeszów
  - Clinical Research Group Sp. Z.O.O, Warsaw
  - High-Med Przychodnia Specjalistycza, Warsaw
  - Centralny Szpital Kliniczny Mswia, Warsaw
- Spain (5):
  - Hospital General Unviersitario de Alicante, Alicante
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital de Manises, Manises
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Data collected through a cut off date of 7 October 2024 have been included in this summary. Participants were enrolled at 52 sites in Argentina, Belgium, Canada, Chile, France, Germany, Italy, Netherlands, Poland, Spain, and the United States.
Groups:
- Vehicle Cream BID to Ruxolitinib 1.5% Cream BID: Participants applied vehicle cream BID through Week 12 to all pruriginous lesions identified at baseline plus an approximate 1 cm area surrounding each lesion in the DBVC Period. At Week 12, the investigator assessed whether the participant required continuation of therapy (IGA-CPG-S score ≥1 and/or the presence of prurigo nodularis-related itching). Those participants who completed 12 weeks of treatment with no safety concerns were eligible to enter the 40-week OLE extension period. Participants randomized to vehicle cream at baseline switched to ruxolitinib 1.5% cream BID and received treatment through Week 52. During the OLE period, participants applied ruxolitinib 1.5% cream BID to prurigo nodularis-affected areas plus an approximate 1 cm area surrounding each pruriginous lesion and/or areas of prurigo nodularis-related itching.
- Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream twice daily (BID) through Week 12 to all pruriginous lesions identified at baseline plus an approximate 1 centimeter (cm) area surrounding each lesion in the Double-blind, Vehicle-controlled (DBVC) Period. At Week 12, the investigator assessed whether the participant required continuation of therapy (Investigator Global Assessment for Stage of Chronic Prurigo [IGA-CPG-S] score ≥1 and/or the presence of prurigo nodularis-related itching). Those participants who completed 12 weeks of treatment with no safety concerns were eligible to enter the 40-week Open-label Extension (OLE) period. Participants randomized to ruxolitinib 1.5% cream at baseline remained on ruxolitinib 1.5% cream BID through Week 52. During the OLE Period, participants applied ruxolitinib 1.5% cream BID to prurigo nodularis-affected areas plus an approximate 1 cm area surrounding each pruriginous lesion and/or areas of prurigo nodularis-related itching.
Period: 12-week DBVC Period
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Started | 103 | 101
Completed | 84 | 90
Not Completed | 19 | 11
Not completed — Adverse Event | 4 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Sponsor Decision | 1 | 0
Period: 40-week OLE Period
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Started | 84 | 90
Completed | 25 | 20
Not Completed | 59 | 70
Not completed — Adverse Event | 0 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 1 | 1
Not completed — Withdrawal by Subject | 6 | 6
Not completed — Sponsor Decision | 3 | 0
Not completed — Did Not Complete Safety Follow-up Period | 0 | 1
Not completed — Ongoing | 46 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID | Total
Number analyzed (Participants) | 103 | 101 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (13.85) | 59.1 (13.78) | 60.1 (13.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 64 | 129
  Male | 38 | 37 | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian | 84 | 87 | 171
  Black or African American | 9 | 7 | 16
  Asian and Others | 9 | 5 | 14
  Missing | 1 | 2 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 18 | 32
  Not Hispanic or Latino | 88 | 80 | 168
  Unknown | 0 | 1 | 1
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: WI-NRS4 Response at Week 12
Description: WI-NRS4 was defined as the percentage of participants achieving a ≥4-point improvement (reduction) in Worst-Itch Numeric Rating Scale (WI-NRS) score from baseline. The WI-NRS is a patient-reported outcome comprised of a single item rated on a scale from 0 ("no itch") to 10 ("worst imaginable itch"). Participants assessed their worst level of prurigo nodularis-related itch during the past 24 hours on a scale of 0 to 10. The WI-NRS score for baseline was determined by averaging the 7 daily WI-NRS scores before Day 1 (i.e., Days -7 to -1) for all by-visit summaries. The by-visit WI-NRS score for post-baseline visits was determined by averaging the 7 daily WI-NRS scores before the visit day. Participants with missing Week 12 data for any reason, including treatment discontinuation (due to development of atopic dermatitis lesions or any other cause), were defined as nonresponders.
Time Frame: Baseline; Week 12
Population: Intent-to-Treat (ITT) Population: all randomized participants. Treatment groups were defined according to the treatment assignment at the time of randomization regardless of the actual study cream the participant might have applied during their participation in the double-blind, vehicle-controlled period. Participants with a baseline ITCH Score ≥4 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
percentage of participants | 20.6 [13.2 to 29.7] | 44.6 [34.7 to 54.8]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test stratified by IGA-CPG-S score (2 or ≥3) and geographic region (North America or outside of North America); Odds Ratio (OR) = 3.09, 95% CI 2-sided [1.659 to 5.744]
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response Rate Difference = 23.90, 95% CI 2-sided [11.42 to 36.39], Standard Deviation 6.372

2. Secondary Outcome: WI-NRS4 Response at Week 4
Description: WI-NRS4 was defined as the percentage of participants achieving a ≥4-point improvement (reduction) in WI-NRS score from baseline. The WI-NRS is a patient-reported outcome comprised of a single item rated on a scale from 0 ("no itch") to 10 ("worst imaginable itch"). Participants assessed their worst level of prurigo nodularis-related itch during the past 24 hours on a scale of 0 to 10. The WI-NRS score for baseline was determined by averaging the 7 daily WI-NRS scores before Day 1 (i.e., Days -7 to -1) for all by-visit summaries. The by-visit WI-NRS score for post-baseline visits was determined by averaging the 7 daily WI-NRS scores before the visit day.
Time Frame: Baseline; Week 4
Population: ITT Population. Participants with a baseline ITCH Score ≥4 were analyzed. Participants with missing Week 4 data for any reason, including treatment discontinuation (due to development of atopic dermatitis lesions or any other cause), were defined as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
percentage of participants | 12.7 [7.0 to 20.8] | 29.7 [21.0 to 39.6]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0034, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.91, 95% CI 2-sided [1.400 to 6.033]
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response Rate Difference = 16.77, 95% CI 2-sided [5.82 to 27.72], Standard Error of Mean 5.587

3. Secondary Outcome: Percentage of Participants With Overall-Treatment Success at Week 12
Description: Overall-Treatment Success was defined as both a WI-NRS4 response and Investigator's Global Assessment for Stage of Chronic Prurigo Treatment Success (IGA-CPG-S-TS). IGA-CPG-S-TS was defined as an IGA-CPG-S score of 0 or 1 with a ≥2 grade improvement from baseline. The IGA-CPG-S is an overall severity rating of chronic prurigo on a scale of 0 to 4: 0, clear (no pruriginous lesions); 1, almost clear (rare palpable pruriginous lesions [approximately 1-5 lesions]); 2, mild (few palpable pruriginous lesions [approximately 6-19 lesions]); 3, moderate (many palpable pruriginous lesions [approximately 20-100 lesions]); 4, severe (abundant palpable pruriginous lesions [over 100 lesions]).
Time Frame: Baseline; Week 12
Population: ITT Population. Participants with missing Week 12 data for any reason, including treatment discontinuation (due to development of atopic dermatitis lesions or any other cause), were defined as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
percentage of participants | 2.9 [0.6 to 8.3] | 11.9 [6.3 to 19.8]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0164, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.46, 95% CI 2-sided [1.206 to 16.485]
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response Rate Difference = 8.75, 95% CI 2-sided [1.71 to 15.79], Standard Error of Mean 3.591

4. Secondary Outcome: Percentage of Participants With IGA-CPG-S-TS at Week 12
Description: IGA-CPG-S-TS was defined as an IGA-CPG-S score of 0 or 1 with a ≥2 grade improvement from baseline. The IGA-CPG-S is an overall severity rating of chronic prurigo on a scale of 0 to 4: 0, clear (no lesions); 1, almost clear (rare palpable pruriginous lesions [approximately 1-5 lesions]); 2, mild (few palpable pruriginous lesions [approximately 6-19 lesions]); 3, moderate (many palpable pruriginous lesions [approximately 20-100 lesions]); 4, severe (abundant palpable pruriginous lesions [over 100 lesions]).
Time Frame: Baseline; Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
percentage of participants | 3.9 [1.1 to 9.6] | 15.8 [9.3 to 24.4]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0048, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 4.67, 95% CI 2-sided [1.486 to 14.647]
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response Rate Difference = 11.66, 95% CI 2-sided [3.71 to 19.62], Standard Error of Mean 4.060

5. Secondary Outcome: WI-NRS4 Response on Day 7
Description: as for outcome 2
Time Frame: Baseline; Day 7
Population: ITT Population. Participants with a baseline ITCH Score ≥4 were analyzed. Participants with missing Day 7 data for any reason, including treatment discontinuation (due to development of atopic dermatitis lesions or any other cause), were defined as nonresponders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
percentage of participants | 8.9 [3.9 to 16.8] | 23.3 [15.1 to 33.4]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0064, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 3.50, 95% CI 2-sided [1.422 to 8.608]
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; Response Rate Difference = 14.35, 95% CI 2-sided [4.54 to 24.17], Standard Error of Mean 5.008

6. Secondary Outcome: DBVC Period: Change From Baseline in WI-NRS Score at Each Post-baseline Visit
Description: The WI-NRS is a patient-reported outcome comprised of a single item rated on a scale from 0 ("no itch") to 10 ("worst imaginable itch"). Participants assessed their worst level of prurigo nodularis-related itch during the past 24 hours on a scale of 0 to 10. The WI-NRS score for baseline was determined by averaging the 7 daily WI-NRS scores before Day 1 (i.e., Days -7 to -1) for all by-visit summaries. The by-visit WI-NRS score for post-baseline visits was determined by averaging the 7 daily WI-NRS scores before the visit day.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
scores on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 96 | 90
  Change from Baseline at Week 2 | -1.08 (0.196) | -2.07 (0.199)
  Change from Baseline at Week 4: number analyzed (Participants) | 94 | 87
  Change from Baseline at Week 4 | -1.52 (0.247) | -2.94 (0.250)
  Change from Baseline at Week 8: number analyzed (Participants) | 77 | 84
  Change from Baseline at Week 8 | -1.89 (0.267) | -3.58 (0.267)
  Change from Baseline at Week 12: number analyzed (Participants) | 81 | 86
  Change from Baseline at Week 12 | -2.13 (0.273) | -3.80 (0.272)
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 2; Test type: Superiority; p = 0.0005, Mixed Model for Repeated Measures (MMRM); MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least squares Mean Difference = -0.99, 95% CI 2-sided [-1.54 to -0.44], Standard Error of Mean 0.280
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -1.42, 95% CI 2-sided [-2.11 to -0.73], Standard Error of Mean 0.352
Statistical Analysis 3: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 8; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -1.69, 95% CI 2-sided [-2.43 to -0.94], Standard Error of Mean 0.378
Statistical Analysis 4: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 12; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -1.67, 95% CI 2-sided [-2.43 to -0.91], Standard Error of Mean 0.386

7. Secondary Outcome: OLE Period: Change From Baseline in WI-NRS Score at Each Post-baseline Visit
Description: as for outcome 6
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population: all participants who applied ruxolitinib 1.5% cream at least once during the OLE Period. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
scores on a scale
  Change from Baseline at Week 14: number analyzed (Participants) | 74 | 81
  Change from Baseline at Week 14 | -3.11 (2.526) | -4.45 (2.679)
  Change from Baseline at Week 16: number analyzed (Participants) | 75 | 74
  Change from Baseline at Week 16 | -3.53 (2.640) | -4.41 (2.742)
  Change from Baseline at Week 20: number analyzed (Participants) | 72 | 70
  Change from Baseline at Week 20 | -4.14 (2.521) | -4.58 (2.701)
  Change from Baseline at Week 24: number analyzed (Participants) | 70 | 74
  Change from Baseline at Week 24 | -4.12 (2.650) | -4.64 (2.543)
  Change from Baseline at Week 28: number analyzed (Participants) | 64 | 67
  Change from Baseline at Week 28 | -4.03 (2.643) | -4.66 (2.614)
  Change from Baseline at Week 32: number analyzed (Participants) | 46 | 49
  Change from Baseline at Week 32 | -4.37 (2.735) | -5.40 (2.538)
  Change from Baseline at Week 36: number analyzed (Participants) | 43 | 40
  Change from Baseline at Week 36 | -4.70 (2.808) | -4.86 (2.784)
  Change from Baseline at Week 40: number analyzed (Participants) | 37 | 29
  Change from Baseline at Week 40 | -4.78 (2.777) | -4.43 (2.794)
  Change from Baseline at Week 44: number analyzed (Participants) | 27 | 25
  Change from Baseline at Week 44 | -5.50 (2.496) | -4.81 (2.538)
  Change from Baseline at Week 48: number analyzed (Participants) | 24 | 19
  Change from Baseline at Week 48 | -5.22 (2.501) | -4.78 (2.914)
  Change from Baseline at Week 52: number analyzed (Participants) | 23 | 19
  Change from Baseline at Week 52 | -5.36 (2.546) | -5.03 (2.548)

8. Secondary Outcome: WI-NRS4 Response at Each Post-baseline Visit
Description: as for outcome 2
Time Frame: Baseline; up to Week 52
Population: ITT Population. Participants with a baseline ITCH Score ≥4 were analyzed. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
percentage of participants
  Week 2: number analyzed (Participants) | 96 | 90
  Week 2 | 5.2 [1.7 to 11.7] | 22.2 [14.1 to 32.2]
  Week 4: number analyzed (Participants) | 94 | 87
  Week 4 | 13.8 [7.6 to 22.5] | 34.5 [24.6 to 45.4]
  Week 8: number analyzed (Participants) | 77 | 84
  Week 8 | 22.1 [13.4 to 33.0] | 48.8 [37.7 to 60.0]
  Week 12: number analyzed (Participants) | 81 | 86
  Week 12 | 25.9 [16.8 to 36.9] | 52.3 [41.3 to 63.2]
  Week 14: number analyzed (Participants) | 74 | 81
  Week 14 | 33.8 [23.2 to 45.7] | 56.8 [45.3 to 67.8]
  Week 16: number analyzed (Participants) | 75 | 74
  Week 16 | 42.7 [31.3 to 54.6] | 56.8 [44.7 to 68.2]
  Week 20: number analyzed (Participants) | 72 | 70
  Week 20 | 54.2 [42.0 to 66.0] | 58.6 [46.2 to 70.2]
  Week 24: number analyzed (Participants) | 70 | 74
  Week 24 | 55.7 [43.3 to 67.6] | 60.8 [48.8 to 72.0]
  Week 28: number analyzed (Participants) | 64 | 67
  Week 28 | 54.7 [41.7 to 67.2] | 64.2 [51.5 to 75.5]
  Week 32: number analyzed (Participants) | 46 | 49
  Week 32 | 58.7 [43.2 to 73.0] | 73.5 [58.9 to 85.1]
  Week 36: number analyzed (Participants) | 43 | 40
  Week 36 | 69.8 [53.9 to 82.8] | 72.5 [56.1 to 85.4]
  Week 40: number analyzed (Participants) | 37 | 29
  Week 40 | 64.9 [47.5 to 79.8] | 62.1 [42.3 to 79.3]
  Week 44: number analyzed (Participants) | 27 | 25
  Week 44 | 77.8 [57.7 to 91.4] | 68.0 [46.5 to 85.1]
  Week 48: number analyzed (Participants) | 24 | 19
  Week 48 | 75.0 [53.3 to 90.2] | 63.2 [38.4 to 83.7]
  Week 52: number analyzed (Participants) | 23 | 19
  Week 52 | 73.9 [51.6 to 89.8] | 73.7 [48.8 to 90.9]

9. Secondary Outcome: Time to ≥2-point Improvement From Baseline in WI-NRS Score
Description: as for outcome 6
Time Frame: Baseline; up to Week 52
Population: ITT Population. Participants with a baseline ITCH Score ≥4 were analyzed. Censored participants were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
days | 13.0 [7.0 to 24.0] | 5.0 [4.0 to 8.0]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p < 0.0001, Log Rank; Log-rank test stratified by randomization stratification factors between treatment and vehicle; Hazard Ratio (HR) = 1.925, 95% CI 2-sided [1.406 to 2.636] — Cox regression model stratified by stratification factors (Baseline IGA 2/3, Region North America/ Outside of North America) was conducted to compare the difference in hazard rate between treatment and vehicle

10. Secondary Outcome: Time to ≥4-point Improvement From Baseline in WI-NRS Score
Description: as for outcome 6
Time Frame: Baseline; up to Week 52
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 102 | 101
days | NA [60.0 to NA] — The median and the upper limit of the confidence interval were not estimable because too few participants had events. | 26.0 [18.0 to 39.0]
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Test type: Superiority; p = 0.0002, Log Rank; Log-rank test stratified by randomization stratification factors between treatment and vehicle; Hazard Ratio (HR) = 2.111, 95% CI 2-sided [1.419 to 3.139] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: DBVC Period: Percentage of Participants With a ≥2-point Improvement (Reduction) in Skin Pain NRS Score From Baseline
Description: Participants assessed their worst level of prurigo nodularis-related skin pain during the past 24 hours on a scale of 0 ("no pain") to 10 ("worse imaginable pain"). The Skin Pain NRS score for baseline was determined by averaging the 7 daily NRS scores before Day 1 (i.e., Days -7 to -1) for all by-visit summaries. The by-visit Skin Pain NRS score for post-baseline visits was determined by averaging the 7 daily NRS scores before the visit day.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Participants with a baseline Skin Pain NRS score ≥2 and available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 94 | 94
percentage of participants
  Week 2: number analyzed (Participants) | 89 | 83
  Week 2 | 20.2 [12.4 to 30.1] | 36.1 [25.9 to 47.4]
  Week 4: number analyzed (Participants) | 88 | 80
  Week 4 | 30.7 [21.3 to 41.4] | 56.3 [44.7 to 67.3]
  Week 8: number analyzed (Participants) | 71 | 77
  Week 8 | 33.8 [23.0 to 46.0] | 64.9 [53.2 to 75.5]
  Week 12: number analyzed (Participants) | 75 | 79
  Week 12 | 45.3 [33.8 to 57.3] | 65.8 [54.3 to 76.1]

12. Secondary Outcome: OLE Period: Percentage of Participants With a ≥2-point Improvement (Reduction) in Skin Pain NRS Score From Baseline
Description: as for outcome 11
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Participants with a baseline Skin Pain NRS score ≥2 and available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 76 | 78
percentage of participants
  Week 14: number analyzed (Participants) | 70 | 75
  Week 14 | 57.1 [44.7 to 68.9] | 77.3 [66.2 to 86.2]
  Week 16: number analyzed (Participants) | 70 | 67
  Week 16 | 68.6 [56.4 to 79.1] | 79.1 [67.4 to 88.1]
  Week 20: number analyzed (Participants) | 66 | 64
  Week 20 | 78.8 [67.0 to 87.9] | 78.1 [66.0 to 87.5]
  Week 24: number analyzed (Participants) | 65 | 68
  Week 24 | 76.9 [64.8 to 86.5] | 80.9 [69.5 to 89.4]
  Week 28: number analyzed (Participants) | 59 | 62
  Week 28 | 72.9 [59.7 to 83.6] | 82.3 [70.5 to 90.8]
  Week 32: number analyzed (Participants) | 41 | 44
  Week 32 | 75.6 [59.7 to 87.6] | 86.4 [72.6 to 94.8]
  Week 36: number analyzed (Participants) | 40 | 37
  Week 36 | 77.5 [61.5 to 89.2] | 83.8 [68.0 to 93.8]
  Week 40: number analyzed (Participants) | 35 | 26
  Week 40 | 85.7 [69.7 to 95.2] | 80.8 [60.6 to 93.4]
  Week 44: number analyzed (Participants) | 25 | 22
  Week 44 | 92.0 [74.0 to 99.0] | 81.8 [59.7 to 94.8]
  Week 48: number analyzed (Participants) | 22 | 17
  Week 48 | 90.9 [70.8 to 98.9] | 76.5 [50.1 to 93.2]
  Week 52: number analyzed (Participants) | 21 | 18
  Week 52 | 90.5 [69.6 to 98.8] | 83.3 [58.6 to 96.4]

13. Secondary Outcome: DBVC Period: Change From Baseline in Skin Pain NRS Score at Each Post-baseline Visit
Description: Participants assessed their worst level of prurigo nodularis-related skin pain during the past 24 hours on a scale of 0 ("no pain") to 10 ("worse imaginable pain"). The Skin Pain NRS score for baseline was determined by averaging the 7 daily NRS scores before Day 1 (i.e., Days -7 to -1) for all by-visit summaries. The by-visit Skin Pain NRS score for post-baseline visits was determined by averaging the 7 daily NRS scores before the visit day. Change from baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Analysis was conducted per the MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit). Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
scores on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 93 | 90
  Change from Baseline at Week 2 | -1.02 (0.187) | -1.70 (0.187)
  Change from Baseline at Week 4: number analyzed (Participants) | 92 | 87
  Change from Baseline at Week 4 | -1.44 (0.242) | -2.58 (0.242)
  Change from Baseline at Week 8: number analyzed (Participants) | 75 | 84
  Change from Baseline at Week 8 | -1.84 (0.265) | -2.94 (0.261)
  Change from Baseline at Week 12: number analyzed (Participants) | 79 | 86
  Change from Baseline at Week 12 | -2.05 (0.276) | -3.19 (0.271)
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 2; Test type: Superiority; p = 0.0111, Mixed Model for Repeated Measures; Least Squares Mean Difference = -0.68, 95% CI 2-sided [-1.20 to -0.16], Standard Error of Mean 0.264
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; p = 0.0010, Mixed Model for Repeated Measures; Least Squares Mean Difference = -1.15, 95% CI 2-sided [-1.82 to -0.47], Standard Error of Mean 0.342
Statistical Analysis 3: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 8; Test type: Superiority; p = 0.0034, Mixed Model for Repeated Measures; Least Squares Mean Difference = -1.10, 95% CI 2-sided [-1.84 to -0.37], Standard Error of Mean 0.372
Statistical Analysis 4: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 12; Test type: Superiority; p = 0.0038, Mixed Model for Repeated Measures; Least Squares Mean Difference = -1.13, 95% CI 2-sided [-1.90 to -0.37], Standard Error of Mean 0.387

14. Secondary Outcome: OLE Period: Change From Baseline in Skin Pain NRS Score at Each Post-baseline Visit
Description: as for outcome 13
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
scores on a scale
  Change from Baseline at Week 14: number analyzed (Participants) | 72 | 81
  Change from Baseline at Week 14 | -2.88 (2.540) | -3.77 (2.736)
  Change from Baseline at Week 16: number analyzed (Participants) | 73 | 74
  Change from Baseline at Week 16 | -3.20 (2.496) | -3.71 (2.730)
  Change from Baseline at Week 20: number analyzed (Participants) | 70 | 70
  Change from Baseline at Week 20 | -3.71 (2.485) | -3.93 (2.831)
  Change from Baseline at Week 24: number analyzed (Participants) | 69 | 74
  Change from Baseline at Week 24 | -3.78 (2.798) | -4.01 (2.852)
  Change from Baseline at Week 28: number analyzed (Participants) | 63 | 67
  Change from Baseline at Week 28 | -3.73 (2.757) | -4.00 (2.693)
  Change from Baseline at Week 32: number analyzed (Participants) | 45 | 49
  Change from Baseline at Week 32 | -3.93 (2.895) | -4.51 (2.799)
  Change from Baseline at Week 36: number analyzed (Participants) | 43 | 40
  Change from Baseline at Week 36 | -4.40 (2.988) | -4.48 (2.739)
  Change from Baseline at Week 40: number analyzed (Participants) | 36 | 29
  Change from Baseline at Week 40 | -4.92 (2.785) | -4.07 (2.663)
  Change from Baseline at Week 44: number analyzed (Participants) | 26 | 25
  Change from Baseline at Week 44 | -5.31 (2.465) | -4.47 (2.703)
  Change from Baseline at Week 48: number analyzed (Participants) | 23 | 19
  Change from Baseline at Week 48 | -5.06 (2.453) | -4.34 (2.702)
  Change from Baseline at Week 52: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52 | -4.95 (2.628) | -4.56 (2.383)

15. Secondary Outcome: Percentage of Participants With IGA-CPG-S-TS at Each Postbaseline Visit
Description: IGA-CPG-S-TS was defined as an IGA-CPG-S score of 0 or 1 with a ≥2 grade improvement from baseline. The IGA-CPG-S is an overall severity rating of chronic prurigo nodularis on a scale of 0 to 4: 0, clear (no lesions); 1, almost clear (rare palpable pruriginous lesions [approximately 1-5 lesions]); 2, mild (few palpable pruriginous lesions [approximately 6-19 lesions]); 3, moderate (many palpable pruriginous lesions [approximately 20-100 lesions]); 4, severe (abundant palpable pruriginous lesions [over 100 lesions]). Participants with missing Week 12 data for any reason, including treatment discontinuation (due to development of atopic dermatitis lesions or any other cause), were defined as nonresponders.
Time Frame: Baseline; up to Week 52
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
percentage of participants
  Week 2: number analyzed (Participants) | 97 | 97
  Week 2 | 1.0 [0.0 to 5.6] | 2.1 [0.3 to 7.3]
  Week 4: number analyzed (Participants) | 94 | 95
  Week 4 | 3.2 [0.7 to 9.0] | 8.4 [3.7 to 15.9]
  Week 8: number analyzed (Participants) | 86 | 90
  Week 8 | 5.8 [1.9 to 13.0] | 15.6 [8.8 to 24.7]
  Week 12: number analyzed (Participants) | 84 | 90
  Week 12 | 4.8 [1.3 to 11.7] | 17.8 [10.5 to 27.3]
  Week 14: number analyzed (Participants) | 79 | 87
  Week 14 | 7.6 [2.8 to 15.8] | 23.0 [14.6 to 33.2]
  Week 16: number analyzed (Participants) | 80 | 84
  Week 16 | 17.5 [9.9 to 27.6] | 29.8 [20.3 to 40.7]
  Week 20: number analyzed (Participants) | 77 | 82
  Week 20 | 22.1 [13.4 to 33.0] | 30.5 [20.8 to 41.6]
  Week 24: number analyzed (Participants) | 76 | 80
  Week 24 | 22.4 [13.6 to 33.4] | 32.5 [22.4 to 43.9]
  Week 28: number analyzed (Participants) | 71 | 74
  Week 28 | 25.4 [15.8 to 37.1] | 32.4 [22.0 to 44.3]
  Week 32: number analyzed (Participants) | 50 | 55
  Week 32 | 32.0 [19.5 to 46.7] | 36.4 [23.8 to 50.4]
  Week 36: number analyzed (Participants) | 44 | 46
  Week 36 | 34.1 [20.5 to 49.9] | 39.1 [25.1 to 54.6]
  Week 40: number analyzed (Participants) | 39 | 35
  Week 40 | 33.3 [19.1 to 50.2] | 40.0 [23.9 to 57.9]
  Week 44: number analyzed (Participants) | 30 | 28
  Week 44 | 43.3 [25.5 to 62.6] | 42.9 [24.5 to 62.8]
  Week 48: number analyzed (Participants) | 25 | 21
  Week 48 | 44.0 [24.4 to 65.1] | 28.6 [11.3 to 52.2]
  Week 52: number analyzed (Participants) | 24 | 20
  Week 52 | 50.0 [29.1 to 70.9] | 40.0 [19.1 to 63.9]

16. Secondary Outcome: Percentage of Participants With a IGA-CPG-A Score of 0 or 1 With ≥2-grade Improvement (Reduction) at Each Post-baseline Visit
Description: The Investigator Global Assessment for Activity of Chronic Prurigo (IGA-CPG-A) is an overall severity rating of chronic prurigo nodularis on a scale of 0 to 4: 0, clear (no pruriginous lesions have excoriations or crusts); 1, almost clear (very small proportion of pruriginous lesions have excoriations or crusts [up to approximately 10% of all pruriginous lesions]); 2, mild (minority of pruriginous lesions have excoriations or crusts [approximately 11%-25% of all pruriginous lesions]); 3, moderate (many pruriginous lesions have excoriations or crusts [approximately 26%-75% of all pruriginous lesions]); 4, severe (majority of pruriginous lesions have excoriations or crusts [approximately 76%-100% of all pruriginous lesions]).
Time Frame: Baseline; up to Week 52
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
percentage of participants
  Week 2: number analyzed (Participants) | 97 | 97
  Week 2 | 1.0 [0.0 to 5.6] | 5.2 [1.7 to 11.6]
  Week 4: number analyzed (Participants) | 94 | 95
  Week 4 | 5.3 [1.7 to 12.0] | 11.6 [5.9 to 19.8]
  Week 8: number analyzed (Participants) | 86 | 90
  Week 8 | 14.0 [7.4 to 23.1] | 24.4 [16.0 to 34.6]
  Week 12: number analyzed (Participants) | 84 | 90
  Week 12 | 10.7 [5.0 to 19.4] | 23.3 [15.1 to 33.4]
  Week 14: number analyzed (Participants) | 79 | 87
  Week 14 | 17.7 [10.0 to 27.9] | 25.3 [16.6 to 35.7]
  Week 16: number analyzed (Participants) | 80 | 84
  Week 16 | 31.3 [21.3 to 42.6] | 34.5 [24.5 to 45.7]
  Week 20: number analyzed (Participants) | 77 | 82
  Week 20 | 26.0 [16.6 to 37.2] | 35.4 [25.1 to 46.7]
  Week 24: number analyzed (Participants) | 76 | 80
  Week 24 | 40.8 [29.6 to 52.7] | 38.8 [28.1 to 50.3]
  Week 28: number analyzed (Participants) | 71 | 74
  Week 28 | 39.4 [28.0 to 51.7] | 37.8 [26.8 to 49.9]
  Week 32: number analyzed (Participants) | 50 | 55
  Week 32 | 36.0 [22.9 to 50.8] | 38.2 [25.4 to 52.3]
  Week 36: number analyzed (Participants) | 44 | 46
  Week 36 | 43.2 [28.3 to 59.0] | 41.3 [27.0 to 56.8]
  Week 40: number analyzed (Participants) | 39 | 35
  Week 40 | 41.0 [25.6 to 57.9] | 37.1 [21.5 to 55.1]
  Week 44: number analyzed (Participants) | 30 | 28
  Week 44 | 53.3 [34.3 to 71.7] | 50.0 [30.6 to 69.4]
  Week 48: number analyzed (Participants) | 25 | 21
  Week 48 | 56.0 [34.9 to 75.6] | 47.6 [25.7 to 70.2]
  Week 52: number analyzed (Participants) | 24 | 20
  Week 52 | 62.5 [40.6 to 81.2] | 55.0 [31.5 to 76.9]

17. Secondary Outcome: DBVC Period: Percentage of Participants With >75% Healed Lesions From Prurigo Activity Score (PAS) at Each Postbaseline Visit
Description: The extent and severity of prurigo nodularis was assessed via the PAS (version 1.2). The first 3 items are descriptive of the type, predominant type, distribution, and quantity of pruriginous lesions. The remaining 2 items of the PAS assess disease activity in terms of percentage (i.e., 0%, 1%-25%, 26%-50%, 51%-75%, and 76%-100%) of pruriginous lesions with excoriations/crusts on top (to reflect active scratching) and the percentage (i.e., 100%, 76%-99%, 51%-75%, 26%-50%, and 0%-25%) of healed pruriginous lesions in order to quantify change of prurigo nodularis skin lesions.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
percentage of participants
  Week 2: number analyzed (Participants) | 97 | 97
  Week 2 | 10.3 [5.1 to 18.1] | 14.4 [8.1 to 23.0]
  Week 4: number analyzed (Participants) | 94 | 95
  Week 4 | 21.3 [13.5 to 30.9] | 26.3 [17.8 to 36.4]
  Week 8: number analyzed (Participants) | 86 | 90
  Week 8 | 23.3 [14.8 to 33.6] | 32.2 [22.8 to 42.9]
  Week 12: number analyzed (Participants) | 84 | 90
  Week 12 | 22.6 [14.2 to 33.0] | 32.2 [22.8 to 42.9]

18. Secondary Outcome: OLE Period: Percentage of Participants With >75% Healed Lesions From PAS at Each Postbaseline Visit
Description: as for outcome 17
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Only participants with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
percentage of participants
  Week 14: number analyzed (Participants) | 79 | 87
  Week 14 | 36.7 [26.1 to 48.3] | 37.9 [27.7 to 49.0]
  Week 16: number analyzed (Participants) | 80 | 84
  Week 16 | 40.0 [29.2 to 51.6] | 45.2 [34.3 to 56.5]
  Week 20: number analyzed (Participants) | 77 | 82
  Week 20 | 45.5 [34.1 to 57.2] | 45.1 [34.1 to 56.5]
  Week 24: number analyzed (Participants) | 76 | 80
  Week 24 | 56.6 [44.7 to 67.9] | 48.8 [37.4 to 60.2]
  Week 28: number analyzed (Participants) | 71 | 74
  Week 28 | 63.4 [51.1 to 74.5] | 45.9 [34.3 to 57.9]
  Week 32: number analyzed (Participants) | 50 | 55
  Week 32 | 64.0 [49.2 to 77.1] | 50.9 [37.1 to 64.6]
  Week 36: number analyzed (Participants) | 44 | 46
  Week 36 | 68.2 [52.4 to 81.4] | 56.5 [41.1 to 71.1]
  Week 40: number analyzed (Participants) | 39 | 35
  Week 40 | 64.1 [47.2 to 78.8] | 57.1 [39.4 to 73.7]
  Week 44: number analyzed (Participants) | 30 | 28
  Week 44 | 73.3 [54.1 to 87.7] | 64.3 [44.1 to 81.4]
  Week 48: number analyzed (Participants) | 25 | 21
  Week 48 | 80.0 [59.3 to 93.2] | 61.9 [38.4 to 81.9]
  Week 52: number analyzed (Participants) | 24 | 20
  Week 52 | 75.0 [53.3 to 90.2] | 60.0 [36.1 to 80.9]

19. Secondary Outcome: DBVC Period: Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Each Post-baseline Visit
Description: The DLQI is a simple, 10-question, validated questionnaire to measure how much the skin problem has affected the participant over the previous 7 days. Each question was scored as: 3 (very much), 2 (a lot), 1 (a little), 0 (not at all or not relevant). The DLQI total score was calculated by summing the score of each question, resulting in a maximum of 30 and a minimum of 0. The higher the score, the more the quality of life was impaired. Total DLQI scores were categorized as follows: 0 to 1 (no effect), 2 to 5 (small effect), 6 to 10 (moderate effect), 11 to 20 (very large effect), and 21 to 30 (extremely large effect). Change from Baseline was calculated as the post-baseline visit minus the baseline visit.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
scores on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2 | -4.47 (0.591) | -4.67 (0.576)
  Change from Baseline at Week 4: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4 | -5.37 (0.661) | -5.71 (0.650)
  Change from Baseline at Week 8: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8 | -5.17 (0.677) | -6.25 (0.661)
  Change from Baseline at Week 12: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12 | -4.65 (0.696) | -6.04 (0.675)
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 2; Test type: Superiority; p = 0.8028, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -0.21, 95% CI 2-sided [-1.84 to 1.42], Standard Error of Mean 0.826
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; p = 0.7151, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -0.34, 95% CI 2-sided [-2.17 to 1.49], Standard Error of Mean 0.928
Statistical Analysis 3: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 8; Test type: Superiority; p = 0.2569, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -1.08, 95% CI 2-sided [-2.95 to 0.79], Standard Error of Mean 0.947
Statistical Analysis 4: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 12; Test type: Superiority; p = 0.1555, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = -1.39, 95% CI 2-sided [-3.30 to 0.53], Standard Error of Mean 0.971

20. Secondary Outcome: OLE Period: Change From Baseline in the DLQI Total Score at Each Post-baseline Visit
Description: as for outcome 19
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
scores on a scale
  Change from Baseline at Week 14: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14 | -7.22 (6.179) | -6.90 (6.097)
  Change from Baseline at Week 16: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16 | -7.27 (6.210) | -7.60 (5.979)
  Change from Baseline at Week 20: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20 | -6.97 (6.158) | -6.98 (6.084)
  Change from Baseline at Week 24: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24 | -6.88 (5.421) | -7.28 (6.088)
  Change from Baseline at Week 28: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28 | -7.29 (6.018) | -7.25 (5.845)
  Change from Baseline at Week 32: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32 | -7.06 (5.363) | -7.79 (6.188)
  Change from Baseline at Week 36: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36 | -6.61 (5.004) | -7.74 (6.207)
  Change from Baseline at Week 40: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40 | -6.62 (4.663) | -6.61 (5.963)
  Change from Baseline at Week 44: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44 | -6.41 (4.179) | -6.56 (5.094)
  Change from Baseline at Week 48: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48 | -4.96 (4.704) | -6.30 (4.846)
  Change from Baseline at Week 52: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52 | -5.95 (4.146) | -6.53 (5.521)

21. Secondary Outcome: DBVC Period: Change From Baseline in European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) Visual Analog Scale (VAS) Score at Each Postbaseline Visit
Description: The EQ-5D-5L is a standardized instrument for use as a measure of health outcome. The EQ-5D-5L consists of 2 sections: the EQ-5D descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 response levels, which are coded by single-digit numbers: 1 = no problems, 2 = slight problems, 3 = moderate problems, 4 = severe problems, 5 = unable to/extreme problems. The EQ VAS records the participant's self-rated health on a vertical VAS (0-100), on which the endpoints are labeled "the best health you can imagine" (100 score) and "the worst health you can imagine" (0 score). Change from Baseline was calculated as the post-baseline value minus the baseline value.
Time Frame: Baseline; up to Week 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
scores on a scale
  Change from Baseline at Week 2: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2 | 3.00 (1.948) | 7.90 (1.896)
  Change from Baseline at Week 4: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4 | 5.59 (1.940) | 8.90 (1.914)
  Change from Baseline at Week 8: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8 | 2.52 (2.189) | 9.83 (2.133)
  Change from Baseline at Week 12: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12 | 5.35 (2.235) | 11.26 (2.171)
Statistical Analysis 1: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 2; Test type: Superiority; p = 0.0736, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = 4.90, 95% CI 2-sided [-0.47 to 10.27], Standard Error of Mean 2.722
Statistical Analysis 2: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 4; Test type: Superiority; p = 0.2265, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = 3.31, 95% CI 2-sided [-2.07 to 8.69], Standard Error of Mean 2.729
Statistical Analysis 3: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 8; Test type: Superiority; p = 0.0180, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = 7.31, 95% CI 2-sided [1.27 to 13.35], Standard Error of Mean 3.061
Statistical Analysis 4: Comparison: Vehicle Cream BID to Ruxolitinib 1.5% Cream BID vs Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID; Week 12; Test type: Superiority; p = 0.0600, Mixed Model for Repeated Measures; MMRM model: (Response Variable = Treatment + Stratification Factors [IGA-CPG-S/Region] + Visit + Treatment*Visit); Least Squares Mean Difference = 5.90, 95% CI 2-sided [-0.25 to 12.06], Standard Error of Mean 3.119

22. Secondary Outcome: OLE Period: Change From Baseline in EQ-5D-5L VAS Score at Each Postbaseline Visit
Description: as for outcome 21
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
scores on a scale
  Change from Baseline at Week 14: number analyzed (Participants) | 76 | 84
  Change from Baseline at Week 14 | 7.54 (19.216) | 10.49 (19.469)
  Change from Baseline at Week 16: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16 | 6.06 (20.263) | 12.06 (18.268)
  Change from Baseline at Week 20: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20 | 8.51 (18.617) | 12.34 (20.446)
  Change from Baseline at Week 24: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24 | 10.12 (17.469) | 11.61 (19.913)
  Change from Baseline at Week 28: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28 | 10.24 (17.467) | 12.86 (19.851)
  Change from Baseline at Week 32: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32 | 8.43 (14.200) | 14.19 (18.760)
  Change from Baseline at Week 36: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36 | 9.85 (15.779) | 13.58 (16.684)
  Change from Baseline at Week 40: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40 | 5.95 (13.603) | 14.94 (16.165)
  Change from Baseline at Week 44: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44 | 6.62 (14.027) | 11.81 (16.948)
  Change from Baseline at Week 48: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48 | 7.33 (14.288) | 6.65 (14.929)
  Change from Baseline at Week 52: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52 | 10.32 (8.676) | 8.89 (11.338)

23. Secondary Outcome: DBVC Period: Change From Baseline in EQ-5D-5L Dimension Scores at Each Postbaseline Visit
Description: as for outcome 21
Time Frame: Baseline; up to Week 12
Population: ITT Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 101
scores on a scale
  Change from Baseline at Week 2, Mobility: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2, Mobility | -0.18 (0.912) | -0.07 (0.606)
  Change from Baseline at Week 4, Mobility: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4, Mobility | -0.21 (0.742) | -0.08 (0.810)
  Change from Baseline at Week 8, Mobility: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8, Mobility | -0.19 (0.813) | -0.08 (0.690)
  Change from Baseline at Week 12, Mobility: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12, Mobility | -0.13 (0.973) | -0.14 (0.714)
  Change from Baseline at Week 2, Self-care: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 2, Self-care | -0.01 (0.533) | -0.05 (0.533)
  Change from Baseline at Week 4, Self-care: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4, Self-care | -0.06 (0.505) | -0.07 (0.493)
  Change from Baseline at Week 8, Self-care: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8, Self-care | -0.06 (0.581) | -0.06 (0.581)
  Change from Baseline at Week 12, Self-care: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12, Self-care | 0.03 (0.636) | -0.06 (0.488)
  Change from Baseline at Week 2, Usual activities: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2, Usual activities | -0.19 (0.782) | -0.25 (0.714)
  Change from Baseline at Week 4, Usual activities: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4, Usual activities | -0.11 (0.785) | -0.21 (0.727)
  Change from Baseline at Week 8, Usual activities: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8, Usual activities | -0.23 (0.811) | -0.22 (0.726)
  Change from Baseline at Week 12, Usual activities: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12, Usual activities | -0.05 (0.727) | -0.27 (0.723)
  Change from Baseline at Week 2, Pain/discomfort: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2, Pain/discomfort | -0.42 (1.136) | -0.56 (0.953)
  Change from Baseline at Week 4, Pain/discomfort: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4, Pain/discomfort | -0.67 (1.132) | -0.67 (1.039)
  Change from Baseline at Week 8, Pain/discomfort: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8, Pain/discomfort | -0.56 (1.112) | -0.66 (1.080)
  Change from Baseline at Week 12, Pain/discomfort: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12, Pain/discomfort | -0.54 (1.078) | -0.70 (1.074)
  Change from Baseline at Week 2, Anxiety/depression: number analyzed (Participants) | 89 | 95
  Change from Baseline at Week 2, Anxiety/depression | -0.20 (1.013) | -0.24 (0.919)
  Change from Baseline at Week 4, Anxiety/depression: number analyzed (Participants) | 90 | 90
  Change from Baseline at Week 4, Anxiety/depression | -0.28 (1.102) | -0.34 (0.996)
  Change from Baseline at Week 8, Anxiety/depression: number analyzed (Participants) | 80 | 86
  Change from Baseline at Week 8, Anxiety/depression | -0.19 (1.045) | -0.37 (0.934)
  Change from Baseline at Week 12, Anxiety/depression: number analyzed (Participants) | 80 | 88
  Change from Baseline at Week 12, Anxiety/depression | -0.24 (1.105) | -0.32 (0.941)

24. Secondary Outcome: OLE Period: Change From Baseline in EQ-5D-5L Dimension Scores at Each Postbaseline Visit
Description: as for outcome 21
Time Frame: Baseline; up to Week 52
Population: Open-label Extension Population. Only participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
scores on a scale
  Change from Baseline at Week 14, Mobility: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14, Mobility | -0.05 (0.728) | -0.10 (0.882)
  Change from Baseline at Week 16, Mobility: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16, Mobility | -0.17 (0.657) | -0.11 (0.786)
  Change from Baseline at Week 20, Mobility: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20, Mobility | -0.22 (0.798) | -0.19 (0.748)
  Change from Baseline at Week 24, Mobility: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24, Mobility | -0.27 (0.886) | -0.12 (0.697)
  Change from Baseline at Week 28, Mobility: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28, Mobility | -0.10 (0.917) | -0.15 (0.856)
  Change from Baseline at Week 32, Mobility: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32, Mobility | -0.09 (0.974) | -0.25 (0.926)
  Change from Baseline at Week 36, Mobility: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36, Mobility | -0.15 (0.963) | -0.16 (0.843)
  Change from Baseline at Week 40, Mobility: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40, Mobility | -0.24 (0.830) | -0.12 (0.740)
  Change from Baseline at Week 44, Mobility: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44, Mobility | -0.14 (0.833) | 0.07 (0.829)
  Change from Baseline at Week 48, Mobility: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48, Mobility | -0.08 (0.974) | -0.05 (0.999)
  Change from Baseline at Week 52, Mobility: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52, Mobility | -0.23 (0.869) | 0.05 (0.970)
  Change from Baseline at Week 14, Self-care: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14, Self-care | 0.04 (0.552) | 0.02 (0.613)
  Change from Baseline at Week 16, Self-care: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16, Self-care | 0.00 (0.562) | -0.11 (0.521)
  Change from Baseline at Week 20, Self-care: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20, Self-care | 0.05 (0.521) | -0.06 (0.486)
  Change from Baseline at Week 24, Self-care: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24, Self-care | -0.04 (0.455) | 0.00 (0.465)
  Change from Baseline at Week 28, Self-care: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28, Self-care | -0.04 (0.438) | -0.10 (0.452)
  Change from Baseline at Week 32, Self-care: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32, Self-care | -0.09 (0.351) | 0.00 (0.280)
  Change from Baseline at Week 36, Self-care: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36, Self-care | -0.05 (0.384) | -0.02 (0.266)
  Change from Baseline at Week 40, Self-care: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40, Self-care | -0.03 (0.287) | 0.00 (0.000)
  Change from Baseline at Week 44, Self-care: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44, Self-care | 0.00 (0.267) | 0.00 (0.277)
  Change from Baseline at Week 48, Self-care: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48, Self-care | -0.04 (0.204) | -0.05 (0.224)
  Change from Baseline at Week 52, Self-care: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52, Self-care | 0.05 (0.375) | -0.05 (0.229)
  Change from Baseline at Week 14, Usual activities: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14, Usual activities | -0.13 (0.838) | -0.22 (0.773)
  Change from Baseline at Week 16, Usual activities: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16, Usual activities | -0.21 (0.800) | -0.28 (0.742)
  Change from Baseline at Week 20, Usual activities: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20, Usual activities | -0.24 (0.791) | -0.31 (0.773)
  Change from Baseline at Week 24, Usual activities: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24, Usual activities | -0.25 (0.813) | -0.21 (0.643)
  Change from Baseline at Week 28, Usual activities: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28, Usual activities | -0.21 (0.783) | -0.32 (0.858)
  Change from Baseline at Week 32, Usual activities: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32, Usual activities | -0.36 (0.735) | -0.33 (0.706)
  Change from Baseline at Week 36, Usual activities: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36, Usual activities | -0.15 (0.654) | -0.28 (0.630)
  Change from Baseline at Week 40, Usual activities: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40, Usual activities | -0.16 (0.602) | -0.18 (0.683)
  Change from Baseline at Week 44, Usual activities: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44, Usual activities | -0.24 (0.425) | -0.11 (0.698)
  Change from Baseline at Week 48, Usual activities: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48, Usual activities | 0.04 (0.550) | -0.20 (0.768)
  Change from Baseline at Week 52, Usual activities: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52, Usual activities | -0.32 (0.568) | -0.11 (0.809)
  Change from Baseline at Week 14, Pain/discomfort: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14, Pain/discomfort | -0.78 (1.040) | -0.67 (1.057)
  Change from Baseline at Week 16, Pain/discomfort: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16, Pain/discomfort | -0.86 (0.969) | -0.73 (1.089)
  Change from Baseline at Week 20, Pain/discomfort: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20, Pain/discomfort | -0.77 (0.915) | -0.68 (1.199)
  Change from Baseline at Week 24, Pain/discomfort: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24, Pain/discomfort | -0.88 (0.897) | -0.81 (1.062)
  Change from Baseline at Week 28, Pain/discomfort: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28, Pain/discomfort | -0.90 (0.964) | -0.83 (0.956)
  Change from Baseline at Week 32, Pain/discomfort: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32, Pain/discomfort | -0.91 (0.929) | -0.92 (1.100)
  Change from Baseline at Week 36, Pain/discomfort: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36, Pain/discomfort | -0.85 (1.062) | -0.95 (1.090)
  Change from Baseline at Week 40, Pain/discomfort: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40, Pain/discomfort | -1.05 (1.104) | -0.85 (1.093)
  Change from Baseline at Week 44, Pain/discomfort: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44, Pain/discomfort | -1.00 (1.000) | -0.78 (1.121)
  Change from Baseline at Week 48, Pain/discomfort: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48, Pain/discomfort | -0.83 (0.963) | -0.80 (1.105)
  Change from Baseline at Week 52, Pain/discomfort: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52, Pain/discomfort | -0.95 (0.999) | -0.84 (1.015)
  Change from Baseline at Week 14, Anxiety/depression: number analyzed (Participants) | 76 | 86
  Change from Baseline at Week 14, Anxiety/depression | -0.25 (1.179) | -0.37 (1.030)
  Change from Baseline at Week 16, Anxiety/depression: number analyzed (Participants) | 77 | 82
  Change from Baseline at Week 16, Anxiety/depression | -0.35 (1.167) | -0.48 (0.972)
  Change from Baseline at Week 20, Anxiety/depression: number analyzed (Participants) | 74 | 80
  Change from Baseline at Week 20, Anxiety/depression | -0.30 (0.961) | -0.38 (0.933)
  Change from Baseline at Week 24, Anxiety/depression: number analyzed (Participants) | 73 | 75
  Change from Baseline at Week 24, Anxiety/depression | -0.30 (0.953) | -0.33 (0.890)
  Change from Baseline at Week 28, Anxiety/depression: number analyzed (Participants) | 68 | 71
  Change from Baseline at Week 28, Anxiety/depression | -0.26 (0.924) | -0.28 (0.897)
  Change from Baseline at Week 32, Anxiety/depression: number analyzed (Participants) | 47 | 52
  Change from Baseline at Week 32, Anxiety/depression | -0.28 (0.800) | -0.38 (0.867)
  Change from Baseline at Week 36, Anxiety/depression: number analyzed (Participants) | 41 | 43
  Change from Baseline at Week 36, Anxiety/depression | -0.17 (0.892) | -0.63 (0.952)
  Change from Baseline at Week 40, Anxiety/depression: number analyzed (Participants) | 37 | 33
  Change from Baseline at Week 40, Anxiety/depression | -0.27 (0.732) | -0.55 (0.905)
  Change from Baseline at Week 44, Anxiety/depression: number analyzed (Participants) | 29 | 27
  Change from Baseline at Week 44, Anxiety/depression | -0.21 (0.940) | -0.33 (1.038)
  Change from Baseline at Week 48, Anxiety/depression: number analyzed (Participants) | 24 | 20
  Change from Baseline at Week 48, Anxiety/depression | -0.04 (0.806) | -0.15 (0.933)
  Change from Baseline at Week 52, Anxiety/depression: number analyzed (Participants) | 22 | 19
  Change from Baseline at Week 52, Anxiety/depression | -0.27 (0.767) | -0.32 (0.749)

25. Secondary Outcome: DBVC Period: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: up to Week 12
Population: Safety Population: all participants who applied ruxolitinib 1.5% cream or vehicle cream at least once. Treatment groups were determined according to the actual treatment the participant applied on Day 1 regardless of assigned treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 100
Participants | 37 | 31

26. Secondary Outcome: DBVC Period: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of TEAEs was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 Grades 1 through 5. The investigator made an assessment of intensity for each TEAE and assigned it to one of the following categories: Grade 1, mild; Grade 2, moderate; Grade 3, severe or medically significant but not immediately life threatening; Grade 4, life-threatening consequences; Grade 5, fatal.
Time Frame: up to Week 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 103 | 100
Participants | 5 | 4

27. Secondary Outcome: OLE Period: Number of Participants With Any TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug.
Time Frame: from beginning of Week 13 up to Week 56
Population: Open-label Extension Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
Participants | 37 | 46

28. Secondary Outcome: OLE Period: Number of Participants With Any ≥Grade 3 TEAE
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered drug related. An AE can therefore have been any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study cream. A TEAE was defined as any AE reported for the first time or the worsening of a pre-existing event after the first application of study drug. The severity of TEAEs was assessed using CTCAE version 5.0 Grades 1 through 5. The investigator made an assessment of intensity for each TEAE and assigned it to one of the following categories: Grade 1, mild; Grade 2, moderate; Grade 3, severe or medically significant but not immediately life threatening; Grade 4, life-threatening consequences; Grade 5, fatal.
Time Frame: from beginning of Week 13 up to Week 56
Population: Open-label Extension Population
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Cream BID to Ruxolitinib 1.5% Cream BID | Ruxolitinib 1.5% Cream BID to Ruxolitinib 1.5% Cream BID
Number analyzed (Participants) | 84 | 90
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: up to Week 56
Description: For participants who were on vehicle up to Week 12 and then switched to ruxolitinib, adverse events are presented by the treatment they were on at the onset of the event. Data have been presented for the Safety Population, comprised of all participants who applied at least one dose of ruxolitinib 1.5% cream or vehicle cream.
Groups:
- Vehicle Cream BID: Participants applied vehicle cream BID through Week 12 to all pruriginous lesions identified at baseline plus an approximate 1 cm area surrounding each lesion in the Double-blind, Vehicle-controlled (DBVC) Period.
- Ruxolitinib 1.5% Cream BID: Participants applied ruxolitinib 1.5% cream BID to all pruriginous lesions identified at baseline plus an approximate 1 centimeter (cm) area surrounding each lesion for 12 weeks in the DBVC Period and for 40 weeks in the OLE Period. Participants who applied matching vehicle cream BID for 12 weeks during the DBVC Period and completed the Week 12 assessments with no safety concerns applied ruxolitinib 1.5% cream for 40 weeks during the OLE Period.
Arm/Group | Vehicle Cream BID | Ruxolitinib 1.5% Cream BID
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/184
Serious Adverse Events (participants affected / at risk) | 5/103 | 13/184
Other Adverse Events (participants affected / at risk) | 6/103 | 27/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=103) | Ruxolitinib 1.5% Cream BID (N=184)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle Cream BID (N=103) | Ruxolitinib 1.5% Cream BID (N=184)
COVID-19 (Infections and infestations) | 4 (4) | 10 (10)
Nasopharyngitis (Infections and infestations) | 2 (2) | 17 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (2):
  • Study Protocol (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/38/NCT05755438/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT05755438/SAP_001.pdf